CLINICAL TRIAL: NCT02440633
Title: A Phase 1,Open -Label Study to Assess the Absorption, Metabolism and Excretion of 14C-OPS-2071 Following a Single Oral Dose to Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 341-14-001
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Bacterial Enteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-OPS-2071 (Experimental): Suspension containing 50 mg of 14C-OPS-2071
  Interventions: Drug: 14C-OPS-2071

INTERVENTIONS:
Drug: 14C-OPS-2071 — Subjects will swallow Single 25 mL of suspension containing 50 mg of 14C-OPS-2071 directly.

SUMMARY:
To obtain absorption, metabolism and excretion data for parent drug and any metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Body mass index (BMI) between 18.5 and 25.0 kg/m2, inclusive
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

* Subjects who have a significant history of alcoholism or drug/chemical abuse, as determined by the Investigator.
* Subjects who smoke, or who have used nicotine within 3 months prior to screening..
* Subjects who have a significant history of drug allergy, as determined by the Investigator.
* Subjects who have any clinically significant abnormal physical examination finding.
* Subjects who have any clinically significant medical history, as determined by the Investigator.
* Subjects who are exposed to radiation as a result of their occupation.
* Subjects who have had an X ray or CT scan, or who have participated in any trial involving a radiolabelled investigational product or have been exposed to radiolabelled substances within 12 months prior to dose administration.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Kotobuki, Study Director — Small Global, Division of New Product Evaluation and Development
Locations (1):
- Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 14C-OPS-2071
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 14C-OPS-2071
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: The Amounts of Radioactivity Excreted in Urine and Faeces
Description: A single dose of 14C-OPS-2071was administered as an oral suspension under fasting conditions on the morning of Day 1. We evaluated the cumulative excretion of total radioactivity (%) in feces and urine, up to 168 hours postdose.
Time Frame: up to144-168h postdose.
Measure: Mean (Standard Deviation); unit: percentage of administered dose
Arm/Group | Feces | Urine | Total
Number analyzed (Participants) | 8 | 8 | 8
percentage of administered dose | 78.0 (13.1) | 6.08 (1.71) | 84.1 (12.7)

2. Primary Outcome: Area Under Curve (AUC) of Total Radioactivity in Plasma and Whole Blood
Description: A single dose of 14C-OPS-2071was administered as an oral suspension under fasting conditions on the morning of Day 1. We measured total radioactivity in plasma and whole blood each. We evaluated AUC 0-168h of total radioactivity in plasma and whole blood each. The AUCs in plasma and whole blood are of total radioactivity including the parent and metabolites.
Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 h postdose.
Measure: Mean (Standard Deviation); unit: μg eq.·h/L
Arm/Group | Plasma | Whole Blood
Number analyzed (Participants) | 8 | 8
μg eq.·h/L | 649.0 (486.0) | 411.0 (73.9)

3. Primary Outcome: AUC of OPS-2071 in Plasma
Description: A single dose of 14C-OPS-2071was administered as an oral suspension under fasting conditions on the morning of Day 1. We measured OPS-2071 concentration in plasma and evaluated AUC 0-168h of OPS-2071 in plasma.
Time Frame: predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 h postdose.
Measure: Mean (Standard Deviation); unit: μg·h/L
Arm/Group | Plasma
Number analyzed (Participants) | 8
μg·h/L | 392.0 (95.8)

ADVERSE EVENTS:
Time Frame: From informed Consent up to 22 days post dose
Arm/Group | 14C-OPS-2071
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14C-OPS-2071 (N=8)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increase (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No